CLINICAL TRIAL: NCT06193863
Title: Special Drug Use Investigation of Rivaroxaban in Pediatric Patients With Congenital Heart Disease (CHD) Who Had Undergone the Fontan Procedure
Brief Title: An Observational Study to Learn More About How Safe Rivaroxaban is And How Well it Works in Children With Congenital Heart Disease Who Had a Heart Surgery Called the Fontan Procedure
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 22468
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Prevention of Venous Thromboembolism; Congenital Heart Disease; Fontan Procedure; Children
Keywords: Prevention of thrombi/emboli formation
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rivaroxaban: Pediatric patients with CHD who had undergone the Fontan procedure were prescribed with Xarelto before enrollment.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — At the discretion of the treating physician, based on the recommendations written in the local product information.

SUMMARY:
This is an observational study in which the data from children with congenital heart disease will be collected and studied. These children will include those who are prescribed rivaroxaban by their doctors after a heart surgery called the Fontan procedure.

Congenital heart disease (CHD) is a heart problem that some children are born with. It sometimes requires a surgery called the Fontan procedure to improve the blood flow in the body. The Fontan procedure can increase the risk of the formation of blood clots in the blood vessels (called thrombosis), which might lead to death.

The study drug, rivaroxaban, is an approved treatment for preventing the formation of blood clots. It is a type of anticoagulant that prevents the blood from clotting by blocking a protein responsible for it. Rivaroxaban can increase the risk of bleeding.

A previous study suggested that the number of major bleeding episodes did not differ much while taking rivaroxaban compared to aspirin in children with CHD who had undergone the Fontan procedure. However, there is limited information available for Japanese patients.

To better understand the safety and potential risks of this drug in children, more knowledge is needed about the use of rivaroxaban in the real world.

The main purpose of this study is to learn more about the occurrence of major bleeding or non-major bleeding in children who were treated with rivaroxaban. Major bleeding is defined as a serious or life-threatening bleeding episode that can have an impact on a person's health and requires medical attention. Non-major bleeding is defined as a type of bleeding that may negatively impact a person's health if not treated.

The data will be collected from December 2023 to June 2026. Researchers will observe each participant for up to 30 days after stopping the treatment or for a maximum of 2 years.

In this study, only available data from regular health visits will be collected. No visits or tests are required as part of this study. Researchers will use the medical records or interview the children and/or their guardians during regular visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the age of 18 years
* Patients diagnosed with CHD who had undergone the Fontan procedure by the investigator under routine clinical practice, and must be judged appropriate for/decided to be treated with rivaroxaban by the investigator under routine clinical practice
* Informed consent form obtained from a legal representative

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice
* Contraindications according to the local marketing authorization
* Previous treatment with rivaroxaban

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under the age of 18 years with a diagnosis of CHD who had undergone the Fontan procedure treated with rivaroxaban has been made by the treating physician before study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of major bleeding or clinically relevant non-major bleeding | Up to 2 years

SECONDARY OUTCOMES:
Occurrence of any bleeding | Up to 2 years
Occurrence of all adverse events (AEs) | Up to 2 years
Occurrence of thrombotic events | Up to 2 years
Descriptive summary of patient demographics/characteristics | Up to 2 years
Dosing patterns of rivaroxaban | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.